CLINICAL TRIAL: NCT00518700
Title: Comfort Evaluation of a New MPS vs. Replenish in Contact Lens Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Innovative medical, Innovative Medical
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 5321
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Corneal Staining

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Other: new MPS
Other: RepleniSH

SUMMARY:
To compare corneal staining after contact lens instillation with a new MPS vs. RepleniSH

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 yrs or older
2. Males or females
3. Any race or ethnic background
4. CL patients using MPS products currently
5. Patients using Contact Lenses habitually (at least 1 month)

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Contact lens use on day of examination.
3. Corneal ectasia.
4. Current use of Restasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milton Hom, OD, FAAO, Principal Investigator — Private Practice
Locations (1):
- Private Practice, Azusa, California, United States